CLINICAL TRIAL: NCT03505229
Title: Stereotactic Body Radiotherapy [SBRT] for High Risk Localised Pancreatic Cancer: a Phase II Study of the Department of Radiation Oncology Royal North Shore Hospital (Span-C - SBRT for Pancreatic Cancer)
Brief Title: Span-C-SBRT for Pancreatic Cancer
Acronym: Span-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Span-C
Record Dates: First submitted 2018-03-05; First posted 2018-04-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: High Risk Localised Pancreatic Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: non randomised-single arm phase II
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): Prior to SBRT, fiducial markers will be placed to aid with image guidance during radiation delivery. Fiducials will be inserted endoscopically (preferable) or intraoperatively. After this procedure, patients will have radiotherapy planning. During treatment, the fiducials will be used for registration with the images acquired during treatment (including kV fluoroscopy, MV or optical). The acquired images may be processed to determine fiducial location using KIM or MATT software from University of Sydney. SBRT 30-45Gray in 5 fractions will be given over 2 weeks.
  Four weeks after completion of SBRT participants will repeat a re-staging PET and CT scans. Those considered to be resectable will proceed to have surgery 6-10 weeks post SBRT.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — Stereotactic Body Radiotherapy (SBRT) 30-45 gray in 5 fractions over 2 weeks will be given to all eligible patients.

SUMMARY:
To assess the freedom from local failure at 12 months after Stereotactic Body Radiotherapy (SBRT). Also to assess the safety, efficacy and feasibility of SBRT in the treatment of high risk localised pancreatic cancer.

DETAILED DESCRIPTION:
Patients must have histologically or cytologically confirmed high risk localised adenocarcinoma of the pancreas, including patients with extrapancreatic extension (Stage IIA), node positive (Stage IIB), borderline resectable or locally advanced pancreatic cancer as defined by Australasian Gastro-Intestinal Trials Group (AGITG) guidelines. ECOG performance status 0-1, suitable for chemotherapy and radiotherapy.

After a minimum of 2 months of neoadjuvant chemotherapy using either an oxaliplatin- based regimen (FOLFOX, FOLFIRINOX, mFOLFIRINOX)+/- immunotherapy/molecular agent or gemcitabine based chemotherapy (eg gemcitabine / gemcitabine/abraxane). Participants will receive SBRT (30-45Gray in 5 fractions over 2 weeks. Prior to SBRT, fiducial markers will be placed to aid with image guidance during radiation delivery. Four weeks after completion of SBRT participants will have re-staging using positron emission tomography (PET) and computed tomography (CT) scan. Participants will be discussed in the multidisciplinary team meeting for consideration of surgery. Those considered to be resectable will proceed to have surgery 6-10 weeks post SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and able to give informed consent
* Patients with histologically or cytologically confirmed locally advanced adenocarcinoma of the pancreas, including patients with extrapancreatic extension (Stage IIA), node positive (Stage IIB), borderline resectable or locally advanced as defined by AGITG guidelines
* ECOG performance status 0-1
* Measurable disease as defined by RECIST 1.1
* Have received or plan to receive chemotherapy
* Successful insertion of fiducial markers

Exclusion Criteria:

* Patients with metastatic pancreas cancer
* Prior abdominal radiotherapy
* Active malignancy excluding non melanomatous skin cancer
* Neuroendocrine pancreatic carcinoma
* Pregnant or lactating women
* Tumour size greater then 70mm
* Age >85

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2028-10-05 (Estimated); Study Completion 2028-10-05 (Estimated)

PRIMARY OUTCOMES:
freedom of local failure | 12 months from end of radiotherapy
  patient who do no have local failure

SECONDARY OUTCOMES:
Incidence of SBRT treatment related adverse events in this group of patients | Acute toxicity-from start of SBRT up to 3 months after SBRT. Late RT toxicity: from 3 months to 2 years after SBRT.
  assess acute and late radiotherapy toxicity using CTCAE version 4.3, to compare toxicity with conventional treatment
Response to neoadjuvant treatments | from date of surgery through to 24 months post surgery
  Determine by pathology and radiological response rates after neoadjuvant treatment,
Feasibility of internal-external correlation model (MATT) | during SBRT radiotherapy treatment
  Determine the feasibility of the University of Sydney internal-external correlation model (MATT) to determine pancreas motion. Feasibility is determined as predicted motion with MATT is within 2mm of actual motion measured with fluoroscopic x-rays of fiducial markers during treatment.
Surgical complications | 30 to 90 days post surgery
  To assess surgical complications
Duration of hospital admission after surgery | from date of surgery through study completion (ie 24 months)
  to assess extended stay in the hospital after surgery
margin negative (R0) resection rate | through study completion, average of 2 years
  to assess margin negative resection rate (i.e. response to treatment)
median overall survival (OS) | 12 months after treatment
  To assess median overall survival after treatment
progression free survival (PFS) | 12 months after treatment
  To assess the PFS rate after treatment
Feasibility of Using Kilovoltage Intra-fraction Monitoring (KIM) to determine pancreas motion | during SBRT radiotherapy treatment
  Determine the feasibility of the University of Sydney Kilovoltage Intra-fraction Monitoring (KIM) software to determine pancreas motion. Feasibility is determined as predicted motion with KIM is within 2mm of actual motion measured with fluoroscopic x-rays of fiducial markers during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: George Hruby, FRANZCR, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
aim to present study data in conferences and medical journals
Supporting Information: CSR
Time Frame: end of trial after analysis

REFERENCES:
- [Derived] Chan J, Kneebone A, Metz G, Booth J, Shepherd M, Kwong C, Brown C, Norton I, Clarke S, Diakos C, Pavlakis N, Mittal A, Samra J, Hruby G. SPAN-C: Results of a Phase II Clinical Trial of Stereotactic Body Radiotherapy in Pancreatic Ductal Adenocarcinoma. J Med Imaging Radiat Oncol. 2025 Aug;69(5):593-600. doi: 10.1111/1754-9485.13874. Epub 2025 Jun 16. PMID 40521621
- [Derived] Madden L, Ahmed A, Stewart M, Chrystall D, Mylonas A, Brown R, Nguyen DT, Keall P, Booth J. CBCT-DRRs superior to CT-DRRs for target-tracking applications for pancreatic SBRT. Biomed Phys Eng Express. 2024 Apr 26;10(3). doi: 10.1088/2057-1976/ad3bb9. PMID 38588646